CLINICAL TRIAL: NCT05804838
Title: Investigation of the Effect of Mindfulness-Based Stress Reduction Program on Depression, Psychological Well-Being and Prenatal Attachment in Pregnant Women
Brief Title: Investigation of the Effect of Mindfulness-Based Stress Reduction Program on in Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ebru Sağıroğlu, Investigator, Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uskudar University ESagiroglu
Record Dates: First submitted 2023-02-24; First posted 2023-04-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Related; Mediation; Depression; Maternal-Fetal Relations
Keywords: depression; conscious awareness; midwifery; prenatal attachment; pregnancy
MeSH Terms: conditions — Negotiating; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled treatments will be carried out in a design. These randomized controlled restrictions should be followed by the Consolidated Standards of Reporting Trials (CONSORT) 2010 guideline controls. The study will consist of an Intervention and a control group.
Masking Description: Since the study is a doctoral thesis, blinding cannot be done due to its nature.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Group (Experimental): Research inclusion criteria
  * Being between 20-35 years old
  * Being her first pregnancy
  * Being between 13 and 24 weeks of gestation
  * Having applied to the pregnant outpatient clinic where the research will be conducted.
  * Not having a hearing-visual impairment
  * Ability to read and write Turkish
  * Volunteering to participate in the research
  * Not having a diagnosis that would constitute an obstacle to physical activity
  * Agreeing to participate in the 8-week MBSR training
  * Being able to use ZOOM Cloud Meetings program
  Interventions: Other: Mindfulness stress reduction program group

INTERVENTIONS:
Other: Mindfulness stress reduction program group — Conscious Awareness Based Stress Reduction program will be applied to women in this group, which will last for 8 weeks. Informed Voluntary Consent Form, Descriptive Characteristics Information Form, Psychological Well-Being Scale, Beck Depression Scale, Prenatal Attachment Scale and Conscious Awareness Scale will be administered to the pregnant women who make up the intervention group before the implementation of the Mindfulness-Based Stress Reduction program. The intervention group will receive 1 session per week. Each session will last 80 minutes. After completing the 8-week MBSR program, data collection forms will be re-applied to the pregnant women in the intervention group and posttest-1 measurements will be made. After the posttest-1 measurements, the pregnants in the intervention group will be given posttest-2 measurements of the pregnants in the intervention group, 1 month after the measurements.

SUMMARY:
This study was planned to examine the effects of the Mindfulness-Based Stress Reduction Program, which is one of the popular concepts of the 21st century, on depression, psychological well-being and prenatal attachment, which are likely to occur as a result of increased stress during an important period that requires adjustment as a result of physical, mental and cognitive changes during pregnancy. It will be conducted in a randomized parallel controlled experimental design type using Consolidated Standards of Reporting Trials (CONSORT) guidelines. It is planned to be carried out with the ZOOM Cloud Meetings program, which is an online education platform, with pregnant women who apply to the Health Sciences University Ümraniye Training and Research Hospital pregnancy polyclinic in the Ümraniye district of Istanbul. The universe of the research will be the pregnant women who applied to the Health Sciences University Ümraniye Training and Research Hospital pregnant outpatient clinic. Primiparous pregnant women who meet the inclusion criteria and willingly agree to participate in the study will be included in the study. 54 people in the intervention group, 54 people in the control group, and a total of 108 people will be taken.

While the Conscious Awareness-Based Stress Reduction Program adapted for pregnant women will be applied to the intervention group, routine follow-up will be applied to the control group within the scope of the outpatient clinic follow-up of the relevant institution. Informed Voluntary Consent Form, Descriptive Characteristics Information Form, Psychological Well-Being Scale, Beck Depression Scale, Prenatal Attachment Scale and Conscious Awareness Scale will be administered to the participants included in the study. As a result of the findings, the discussion and results of the study will be written.

DETAILED DESCRIPTION:
Studies with a high level of evidence evaluating the effectiveness of mindfulness-based practices in obstetrics are limited. It is stated that little is known about the effects of mindfulness-based interventions, which is one of the non-pharmacological methods in the prenatal period, on pregnant women. In a limited number of studies, it is noted that mindfulness-based approaches used in the prenatal period increase the level of awareness by reducing depression, anxiety and anxiety levels. Studies on how to improve the importance of depression, psychological well-being and the bond established with the fetus during pregnancy have been limited to routine birth preparation trainings.

With the importance of living in the moment, focusing on the moment and staying in the moment in the 21st century, mindfulness programs increase the quality of instant life. Especially during the pregnancy period, where many changes are experienced, the studies that adapted the Mindfulness-Based Stress Reduction Program were quite inadequate.

In the literature, many mindfulness-based programs, including the mindfulness-based stress reduction program, have been used in health areas outside the field of midwifery and evidence-based benefits have been demonstrated. However, there is no study examining depression, psychological well-being, and prenatal attachment levels with mindfulness-based stress reduction. The design of the study gives originality to the study with this aspect. In line with the results of the research, in case of methods/methods with which depression, psychological well-being and prenatal attachment efficiency can be determined during pregnancy, compliance with the pregnancy process, reduction in pregnancy complaints, less need for medical intervention and increase in the number of spontaneous vaginal deliveries in line with the preference of the woman in the delivery room, postpartum mother-infant attachment, Considering that there will be an increase in compliance with the breastfeeding process and newborn care, it can be presented as an alternative method in pregnant training in the preparation process for childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-35 years old
* Being her first pregnancy
* Being between 13 and 24 weeks of gestation
* Having applied to the pregnant outpatient clinic where the research will be conducted.
* Not having a hearing-visual impairment
* Ability to read and write Turkish
* Volunteering to participate in the research
* Not having a diagnosis that would constitute a physical activity disability.
* Agreeing to participate in the 8-week MBSR training
* Being able to use ZOOM Cloud Meetings program

Exclusion Criteria:

* Being diagnosed with acute/chronic disease during pregnancy
* Having a diagnosis of mental illness in the pregnant
* Multiple pregnancy
* Having participated in any awareness-based training program in the last 1 year

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — being a pregnant woman
Enrollment: 108 (Estimated)
Dates: Start 2024-09-11 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Psychological well-being scale | at inclusion
  The reliability study, the cronbach alpha coefficient was determined as .80. Its consists of a single sub-dimension and 8 items. The items of the scale consist of an answer scale of (1) Strongly disagree, (2) Disagree, (3) Slightly disagree, (4) Undecided, (5) Slightly Agree, (6) Agree, (7) Strongly Agree.
  All items of the scale are expressed positively. The scores that can be obtained from the scale range from 8 to 56, and it is stated that the person with a high score has a certain psychological resource and power.
  The application time for each pregnant takes approximately 5 minutes.
Beck depression scale | at inclusion
  This scale is a 21-item self-assessment scale and measures depressive symptoms and characteristic approaches.
  It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. Each item was given a score between 0 and 3, and the highest score that could be obtained from the scale was calculated as 63 and the lowest score as 0.
  A high score on the scale indicates that the severity or level of depression is high.
  The application time for each pregnant takes approximately 20 minutes.
Prenatal attachment scale | at inclusion
  It is a 15-item scale. High scores on the scale indicate high conscious awareness. It is a 6-point Likert-type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The application time for each pregnant takes approximately 25 minutes.
Conscious awareness scale | at inclusion
  Scale is a 15-item scale that measures the general tendency to be aware of and attentive to momentary experiences in daily life.
  The Conscious Awareness Scale has a single factor structure and gives a single total score.
  High scores on the scale indicate high conscious awareness. The Conscious Awareness Scale is a 6-point Likert type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The validity and reliability results of the Conscious Awareness Scale have shown that the Conscious Awareness Scale is a highly valid and reliable measurement tool.
  The internal consistency coefficient (coefficient alpha) of the scale is 0.82. The application time for each pregnant takes approximately 10 minutes.

SECONDARY OUTCOMES:
Psychological well-being scale | At the end of the Mindfulness-Based Stress Reduction Program (week 8)
  The reliability study, the cronbach alpha coefficient was determined as .80. Its consists of a single sub-dimension and 8 items. The items of the scale consist of an answer scale of (1) Strongly disagree, (2) Disagree, (3) Slightly disagree, (4) Undecided, (5) Slightly Agree, (6) Agree, (7) Strongly Agree.
  All items of the scale are expressed positively. The scores that can be obtained from the scale range from 8 to 56, and it is stated that the person with a high score has a certain psychological resource and power.
  The application time for each pregnant takes approximately 5 minutes.
Beck depression scale | At the end of the Mindfulness-Based Stress Reduction Program (week 8)
  This scale is a 21-item self-assessment scale and measures depressive symptoms and characteristic approaches.
  It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. Each item was given a score between 0 and 3, and the highest score that could be obtained from the scale was calculated as 63 and the lowest score as 0.
  A high score on the scale indicates that the severity or level of depression is high.
  The application time for each pregnant takes approximately 20 minutes.
Prenatal attachment scale | At the end of the Mindfulness-Based Stress Reduction Program (week 8)
  It is a 15-item scale. High scores on the scale indicate high conscious awareness. It is a 6-point Likert-type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The application time for each pregnant takes approximately 25 minutes.
Conscious awareness scale | At the end of the Mindfulness-Based Stress Reduction Program (week 8)
  Scale is a 15-item scale that measures the general tendency to be aware of and attentive to momentary experiences in daily life.
  The Conscious Awareness Scale has a single factor structure and gives a single total score.
  High scores on the scale indicate high conscious awareness. The Conscious Awareness Scale is a 6-point Likert type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The validity and reliability results of the Conscious Awareness Scale have shown that the Conscious Awareness Scale is a highly valid and reliable measurement tool.
  The internal consistency coefficient (coefficient alpha) of the scale is 0.82. The application time for each pregnant takes approximately 10 minutes.

OTHER OUTCOMES:
Psychological well-being scale | At the end of the Mindfulness-Based Stress Reduction Program (at week 12)
  The reliability study, the cronbach alpha coefficient was determined as .80. Its consists of a single sub-dimension and 8 items. The items of the scale consist of an answer scale of (1) Strongly disagree, (2) Disagree, (3) Slightly disagree, (4) Undecided, (5) Slightly Agree, (6) Agree, (7) Strongly Agree.
  All items of the scale are expressed positively. The scores that can be obtained from the scale range from 8 to 56, and it is stated that the person with a high score has a certain psychological resource and power.
  The application time for each pregnant takes approximately 5 minutes.
Beck depression scale | At the end of the Mindfulness-Based Stress Reduction Program (at week 12)
  This scale is a 21-item self-assessment scale and measures depressive symptoms and characteristic approaches.
  It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. Each item was given a score between 0 and 3, and the highest score that could be obtained from the scale was calculated as 63 and the lowest score as 0.
  A high score on the scale indicates that the severity or level of depression is high.
  The application time for each pregnant takes approximately 20 minutes.
Prenatal attachment scale | At the end of the Mindfulness-Based Stress Reduction Program (at week 12)
  It is a 15-item scale. High scores on the scale indicate high conscious awareness. It is a 6-point Likert-type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The application time for each pregnant takes approximately 25 minutes.
Conscious awareness scale | At the end of the Mindfulness-Based Stress Reduction Program (at week 12)
  Scale is a 15-item scale that measures the general tendency to be aware of and attentive to momentary experiences in daily life.
  The Conscious Awareness Scale has a single factor structure and gives a single total score.
  High scores on the scale indicate high conscious awareness. The Conscious Awareness Scale is a 6-point Likert type scale (almost always, often, sometimes, rarely, quite rarely, almost never).
  The validity and reliability results of the Conscious Awareness Scale have shown that the Conscious Awareness Scale is a highly valid and reliable measurement tool.
  The internal consistency coefficient (coefficient alpha) of the scale is 0.82. The application time for each pregnant takes approximately 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Aydın Kartal, Ass.Prof.Dr, Study Director — Saglik Bilimleri Universitesi; Ebru Sağıroğlu, PhD.Stu., Principal Investigator — Uskudar University
Locations (1):
- Istanbul Provincial Health Directorate Umraniye Training and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No